CLINICAL TRIAL: NCT00918671
Title: Treatment of Medication-overuse Headache: 4 Years Follow up
Brief Title: Medication-overuse Headache: 4 Years Follow up
Acronym: MOHfollowup
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2007.2192; 4.2007.2192; 07/4471; 17429
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Medication Overuse Headache
Keywords: Headache; Medication overuse; chronic; relapse
MeSH Terms: conditions — Headache Disorders, Secondary; Headache; Prescription Drug Overuse; Bronchiolitis Obliterans Syndrome; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Medication-overuse headache: Chronic daily headache combined with medication overuse
  Interventions: Other: No new specific intervention

INTERVENTIONS:
Other: No new specific intervention — No new specific intervention

SUMMARY:
From 1 January 2004 to 31 December 2006 64 individuals with probable medication overuse headache were included in a randomized, 1-year open-labeled, multicentre study to evaluate the effect of early introduction of prophylactic treatment compared to abrupt withdrawal and with a control group (ClinicalTrials.gov number NCT00159588). In this follow-up, randomized patients still alive 4 years after primary inclusion time will be invited to a follow up interview, evaluating the headache complaints and the proportion of recurrent medication overuse.

DETAILED DESCRIPTION:
The participants will be interviewed by telephone or consult the study doctor completing a headache diary for at least 1 month before attending the visit.

ELIGIBILITY:
Inclusion Criteria:

* Randomized during the initial trial during 2004-2006.

Ages: 22 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 years remitted to the out-patient clinics of the neuroloical departments of five University Hospitals in Norway with probable medication overuse headache included in a 1-year open-labeled trial during 2004-2006.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Hagen, MD, PhD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Norwegian National headache Centre, NTNU, Trondheim, Norway

REFERENCES:
- [Background] Hagen K, Albretsen C, Vilming ST, Salvesen R, Gronning M, Helde G, Gravdahl G, Zwart JA, Stovner LJ. Management of medication overuse headache: 1-year randomized multicentre open-label trial. Cephalalgia. 2009 Feb;29(2):221-32. doi: 10.1111/j.1468-2982.2008.01711.x. Epub 2008 Sep 24. PMID 18823363
- [Result] Hagen K, Albretsen C, Vilming ST, Salvesen R, Gronning M, Helde G, Gravdahl G, Zwart JA, Stovner LJ. A 4-year follow-up of patients with medication-overuse headache previously included in a randomized multicentre study. J Headache Pain. 2011 Jun;12(3):315-22. doi: 10.1007/s10194-010-0285-1. Epub 2011 Jan 5. PMID 21207237
- [Result] Hagen K, Stovner LJ. A randomized controlled trial on medication-overuse headache: outcome after 1 and 4 years. Acta Neurol Scand Suppl. 2011;(191):38-43. doi: 10.1111/j.1600-0404.2011.01542.x. PMID 21711255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion during the period between January 2008 and May 2010
Pre-assignment Details: Invited to visit a neurologist, interviewed by telephone, give response by letter, or had headache data available in their hospital records
Period: Overall Study
Arm/Group | Medication-overuse Headache
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medication-overuse Headache
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Headache Days/Month After 4 Years Compared to Baseline
Description: Change in headache days/month after 4 years compared to baseline
Time Frame: Baseline and after 4 years
Measure: Mean (Standard Deviation); unit: headache days/month
Arm/Group | Medication-overuse Headache
Number analyzed (Participants) | 60
headache days/month | 6.6 (9.87)

2. Secondary Outcome: Change of Medication Days/Month Compared to Baseline
Time Frame: Baseline and after 4 years' of follow-up
Measure: Mean (Standard Deviation); unit: medication days/month
Arm/Group | Medication-overuse Headache
Number analyzed (Participants) | 60
medication days/month | 9.53 (9.99)

ADVERSE EVENTS:
Arm/Group | Medication-overuse Headache
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No